CLINICAL TRIAL: NCT03936205
Title: Does the Addition of Dexmedetomidine to Morphine Improve the Treatment of Pain in Patients With Metastatic Cancer? A Pilot Study
Brief Title: Dexmedetomidine Addition to Morphine in Patients With Metastatic Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hotel Dieu de France Hospital (Other)
Responsible Party: Principal Investigator, Nicole Naccache, Assistant professor, Hotel Dieu de France Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: FM315
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Refractory Pain; Metastatic Cancer
MeSH Terms: conditions — Pain, Intractable; Neoplasm Metastasis | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Patients allocated to this group receive a combination of Morphine and Dexmedetomidine
  Arms: Dexmedetomidine

SUMMARY:
Pain is a common symptom in patients nearing the end of life. Its prevalence varies between 30 and 75%. Nowadays, morphine is the most used molecule as first line treatment of moderate to severe pain. However, this molecule, considering its side effects, may contribute in part to the discomfort of these patients and may increase the pre-existing agitation or delirium. There is therefore a need to find new agents, other than morphine, for pain control at the end of life, without the limitations that the morphine molecule has. The author reviewed the literature on the role of dexmedetomidine in the treatment of refractory symptoms in palliative care, including pain. It is an agonist of the adrenergic alpha 2 receptor having a sedative, analgesic action and a morphine sparing effect demonstrated postoperatively.

This study aims primarily at demonstrating that dexmedetomidine has a beneficial role in the treatment of pain in patients with metastatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Any painful patient with metastatic cancer
* Whatever type of pain: nociceptive, neuropathic, or mixed
* Age > 18 and <75 years
* Patient under analgesic Tier III treatment: with moderate to severe pain and not relieved by non-opioid conventional treatment
* Patient cooperating capable of responding to the pain assessment by providing a number from 0 to 10 at the VAS
* Patient providing his explicit consent to participate in the study before inclusion (regardless of his inclusion in C or D Group)
* Patients with systolic blood pressure (SBP) ≥ 100 mmHg and a diastolic blood pressure (DBP) ≥ 50 mmHg
* Patients with a heart rate ≥ 50/min

Exclusion Criteria:

* Patient refusal to participate in the study or patient unable to give consent
* Age <18 or > 75 years
* Comatose uncooperative patient unable to respond to the assessment of pain by VAS
* Hypotensive patients with SBP < 100 mmHg and DBP < 60 mmHg or bradycardic with a heart rate < 50/min
* Patient with a heart rhythm disorder, or a disorder of the atrial-ventricular conduction
* Patients under beta-blocker
* Patient with heart failure with an ejection fraction < 40%
* Patient suffering from allergy or previous intolerance to morphine or dexmedetomidine
* Patient with renal impairment with a creatinine clearance <3 0ml/min/1.73m2, or patient under hemodialysis or peritoneal dialysis.
* Patient with severe hepatic impairment with Child-Pugh score at C.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Pain score | 48 hours
  The visual analogue score is used to asses for pain score, the scale varies between 0 and 10 where 0 is no pain and 10 is worst pain encountered
Morphine consumption | 48 hours